CLINICAL TRIAL: NCT06117462
Title: Frailty in Critical Care Unit's Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Mostafa ibrahim sultan, Principle investigator , Residant doctor ,critical care unit ,internal medicine department, Assiut University
Other Study IDs: Fraility in CCU
Record Dates: First submitted 2023-09-28; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: CFS

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Age above 60 eldery: group will be assessed using the Clinical Frailty Scale (CFS) giving patients who are very fit score one and those who are terminally ill score nine.
  Interventions: Other: Assesment of CFS
- age between 18:60 young: group will be assessed using the Clinical Frailty Scale (CFS) giving patients who are very fit score one and those who are terminally ill score nine.
  Interventions: Other: Assesment of CFS

INTERVENTIONS:
Other: Assesment of CFS — Assesment of CFS

SUMMARY:
In the study ,investigator aim to evaluate the frailty syndrome in critically ill patients, in both young and old populations,to determine its imapct on outcome, and impact of ICU in fraility

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients >18 years

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial clinical data will include socio-demographic data, comorbidities (diabetes mellitus (DM), hypertension (HTN), ischemic heart disease (IHD), chronic kidney disease (CKD), chronic liver disease, chronic pulmonary disease, or malignancy), in addition to the acute insult causing the admission.
  Candidates will be divided into two groups, group (A): >60 years, and group (B) aged between 18-60 years, both groups will be assessed using the Clinical Frailty Scale (CFS) giving patients who are very fit score one and those who are terminally ill score nine.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
detect the impact of frailty on outcome(hospital stay and mortality).In Critical care units patients. | the CFS before hospital admission and at day up to 1 week of discharge from CCU, CFS mininum 1 ,maximum 9 patient's basal score[ pre intervention] on day of admission and the outcome score at day of discharge [5day],score 1better than higher
  evaluate the frailty syndrome in critical care unit ,in young and old populations.CFS will report patient's basal score[ pre intervention] on day of admission and the outcome score at day of discharge [5day],score 1better than higher

REFERENCES:
- [Background] Liu Z, Kuo PL, Horvath S, Crimmins E, Ferrucci L, Levine M. A new aging measure captures morbidity and mortality risk across diverse subpopulations from NHANES IV: A cohort study. PLoS Med. 2018 Dec 31;15(12):e1002718. doi: 10.1371/journal.pmed.1002718. eCollection 2018 Dec. PMID 30596641
- [Background] de Rooij SE, Govers A, Korevaar JC, Abu-Hanna A, Levi M, de Jonge E. Short-term and long-term mortality in very elderly patients admitted to an intensive care unit. Intensive Care Med. 2006 Jul;32(7):1039-44. doi: 10.1007/s00134-006-0171-0. Epub 2006 May 9. PMID 16791666
- [Background] Guidet B, de Lange DW, Boumendil A, Leaver S, Watson X, Boulanger C, Szczeklik W, Artigas A, Morandi A, Andersen F, Zafeiridis T, Jung C, Moreno R, Walther S, Oeyen S, Schefold JC, Cecconi M, Marsh B, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Flaatten H; VIP2 study group. The contribution of frailty, cognition, activity of daily life and comorbidities on outcome in acutely admitted patients over 80 years in European ICUs: the VIP2 study. Intensive Care Med. 2020 Jan;46(1):57-69. doi: 10.1007/s00134-019-05853-1. Epub 2019 Nov 29. PMID 31784798
- [Background] Darvall JN, Bellomo R, Bailey M, Young PJ, Rockwood K, Pilcher D. Impact of frailty on persistent critical illness: a population-based cohort study. Intensive Care Med. 2022 Mar;48(3):343-351. doi: 10.1007/s00134-022-06617-0. Epub 2022 Feb 4. PMID 35119497
- [Background] Muscedere J, Waters B, Varambally A, Bagshaw SM, Boyd JG, Maslove D, Sibley S, Rockwood K. The impact of frailty on intensive care unit outcomes: a systematic review and meta-analysis. Intensive Care Med. 2017 Aug;43(8):1105-1122. doi: 10.1007/s00134-017-4867-0. Epub 2017 Jul 4. PMID 28676896